CLINICAL TRIAL: NCT06190873
Title: Effect of Telephone Training on Fear of Movement and Quality of Life in Patients With Lumbar Disc Herniation Surgery: Randomized Controlled Study.
Brief Title: The Effect of Telephone Education on Fear of Movement and Quality of Life in Patients With Lumbar Disc Herniation Surgery.
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Çanakkale Onsekiz Mart University (Other)
Responsible Party: Principal Investigator, Nilgün Temel, graduate student, Çanakkale Onsekiz Mart University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: COMÜ- SBF-NT-01
Record Dates: First submitted 2023-12-11; First posted 2024-01-05 (Actual); Last update posted 2024-01-05 (Actual); Status verified 2023-12

CONDITIONS: Spine Disease; Spinal Deformity
Keywords: life quality; telehealty; tele nursing; kinezyofobi
MeSH Terms: conditions — Spinal Diseases | interventions — Nursing Education Research

STUDY DESIGN:
Intervention Model Description: There will be two groups, one is the control group and the other is the intervention group.
Who Masked: Participant, Outcomes Assessor
Masking Description: Participants will not know which group they belong to.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- group to be trained over the phone (Experimental): This group will be trained by phone for 6 weeks after discharge.
  Interventions: Behavioral: post-discharge rehabilitation training
- Group without telephone training (No Intervention): This group will be given training during their stay in the hospital. There will be no training over the phone after discharge.

INTERVENTIONS:
Behavioral: post-discharge rehabilitation training — Telephone training will be provided for post-discharge rehabilitation
  Other Names: nursingcare; nursing education
  Arms: group to be trained over the phone

SUMMARY:
The aim is to quantify the fear of movement and quality of life of telephone education on lumbar disc herniation surgery.

DETAILED DESCRIPTION:
In the randomized controlled study, patients will be randomized into two categories: experimental and control groups. The experimental group will receive intervention via online information for 6 weeks after discharge. The control group will not be given online training other than standard nursing care. At the end of 6 weeks, the difference between fear of movement and quality of life between the two groups will be examined.

ELIGIBILITY:
Inclusion Criteria:

* being over 18 years old
* knowing how to read and write Turkish
* No hearing or speech impairment
* Having lumbar disc herniation surgery for the first time
* having a personal cell phone
* being discharged 5 days after surgery

Exclusion Criteria:

* being under 18 years old
* being illiterate
* having a hearing and speech disability
* not having a personal cell phone
* staying in the hospital for more than 5 days after surgery

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2023-12-01 (Actual); Primary Completion 2025-01-01 (Estimated); Study Completion 2025-01-01 (Estimated)

PRIMARY OUTCOMES:
movement fear scale | six week
  In the measurement to be made with a four-point Likert type scale, 17 is the lowest score and 68 is the highest score. The higher the score the patient receives, the greater the fear of movement.

SECONDARY OUTCOMES:
quality of life scale | six week
  The score obtained from the scale varies between 0 and 100. As the score obtained from the scale increases, the patient's quality of life increases.

CONTACTS AND LOCATIONS:
Locations (1):
- Çanakkale Mehmet Akif Ersoy Devlet Hastenesi, Çanakkale, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No